CLINICAL TRIAL: NCT06143878
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled and Deucravacitinib Active Comparator-controlled Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of JNJ-77242113 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSO3002; 77242113PSO3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JNJ-77242113 (Experimental): Participants will receive JNJ-77242113 from Week 0 through Week 156 and deucravacitinib matching placebo from Week 0 through Week 24.
  Interventions: Drug: JNJ-77242113; Drug: Deucravacitinib Matching Placebo
- Placebo (Placebo Comparator): Participants will receive matching placebo for JNJ-77242113 from Week 0 through Week 16, matching placebo for deucravacitinib from Week 0 through Week 24 and JNJ-77242113 from Week 16 through Week 156.
  Interventions: Drug: JNJ-77242113; Drug: JNJ-77242113 Matching Placebo; Drug: Deucravacitinib Matching Placebo
- Deucravacitinib (Active Comparator): Participants will receive deucravacitinib from Week 0 through Week 24 and matching placebo for JNJ-77242113 from Week 0 through Week 24 and JNJ-77242113 from Week 24 through Week 156.
  Interventions: Drug: JNJ-77242113; Drug: JNJ-77242113 Matching Placebo; Drug: Deucravacitinib

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally.
Drug: JNJ-77242113 Matching Placebo — JNJ-77242113 matching placebo will be administered orally.
  Arms: Deucravacitinib; Placebo
Drug: Deucravacitinib — Deucravacitinib will be administered orally.
  Arms: Deucravacitinib
Drug: Deucravacitinib Matching Placebo — Deucravacitinib matching placebo will be administered orally.
  Arms: JNJ-77242113; Placebo

SUMMARY:
The purpose of the study is to see how effective JNJ-77242113 is in participants with moderate to severe plaque psoriasis compared to placebo and deucravacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis, with or without psoriatic arthritis (PsA), for at least 26 weeks prior to the first administration of study intervention
* Total body surface area (BSA) greater than or equal to (>=)10 percent (%) at screening and baseline
* Total psoriasis area and severity index (PASI) >=12 at screening and baseline
* Total investigator global assessment (IGA) >=3 at screening and baseline
* Candidate for phototherapy or systemic treatment for plaque psoriasis

Exclusion Criteria:

* Nonplaque form of psoriasis (for example, erythrodermic, guttate, or pustular)
* Current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* A current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, liver, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113, deucravacitinib, or to any of the excipients or components of the study intervention
* Major surgical procedure, (for example, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from surgical procedure, or has a surgical procedure planned during the time the participant is expected to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 or 1 and Greater Than or Equal to (>=) 2-Grade Improvement From Baseline to Week 16 | Baseline and Week 16
  Percentage of participants who achieve an IGA score of 0 or 1 and >=2-Grade improvement from baseline to Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Baseline and Week 16
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving an IGA Score of 0 at Week 16 | Week 16
  Percentage of participants who achieve an IGA score of 0 at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving PASI 75 Response From Baseline to Weeks 4 and 16 | Baseline, Week 4, and Week 16
  Percentage of participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Weeks 4 and 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving PASI 90 Response at Week 8 | Baseline and Week 8
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 8 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving PASI 100 Response at Week 16 | Baseline and Week 16
  Percentage of participants achieving PASI 100 response (100% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Scalp-specific Investigator Global Assessment (ss-IGA) Score of 0 or 1 and >=2 Grade Improvement From Baseline at Week 16 | Baseline and Week 16
  Percentage of participants achieving ss-IGA score of 0 or 1 and >=2 grade improvement from baseline to Week 16 will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Psoriasis Symptom and Signs Diary (PSSD) Symptom Score of 0 at Weeks 8 and 16 | Weeks 8 and 16
  Percentage of participants achieving PSSD symptom score of 0 at Weeks 8 and 16 will be reported. The PSSD includes patient-reported outcome (PRO) questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving >=4 Point Improvement From Baseline in PSSD Itch Score at Weeks 4 and 16 | Baseline, Week 4, and Week 16
  Percentage of participants achieving >=4 Point improvement from baseline in PSSD itch score at Weeks 4 and 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving an IGA Score of 0 or 1 and >=2 Grade Improvement From Baseline at Weeks 16 and 24 | Baseline, Week 16, and Week 24
  Percentage of participants who achieve an IGA score of 0 or 1 and >=2 grade improvement from baseline at Weeks 16 and 24 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving an IGA Score of 0 at Weeks 16 and 24 | Weeks 16 and 24
  Percentage of participants who achieve an IGA score of 0 at Weeks 16 and 24 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving PASI 75 Response at Weeks 16 and 24 | Baseline, Week 16 and Week 24
  Percentage of participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Weeks 16 and 24 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving PASI 90 Response at Weeks 16 and 24 | Baseline, Week 16, and Week 24
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Weeks 16 and 24 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving PASI 100 Response at Weeks 16 and 24 | Baseline, Week 16, and Week 24
  Percentage of participants achieving PASI 100 response (100% improvement in PASI from baseline) at Weeks 16 and 24 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants With PSSD Symptom Score of 0 at Week 16 | Week 16
  Percentage of participants achieving PSSD symptom score 0 at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Number of Participants with Adverse Events (AEs) | Up to 165 weeks
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Serious Adverse Events (SAEs) | Up to 165 weeks
  SAEs are any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, or is medically important.
Change From Baseline in Body Surface Area (BSA) at Week 16 | Baseline and Week 16
  Change from baseline in BSA at Week 16 will be reported. BSA is a commonly used measure of extent of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed (that is, plaque psoriasis).
Change from Baseline in PASI Total Score at Week 16 | Baseline and Week 16
  Change from baseline in PASI total score at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas are assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percent Improvement in PASI Score From Baseline at Week 16 | Baseline and Week 16
  Percent improvement in PASI score from Baseline at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving a Static Physician's Global Assessment of Genitalia (sPGA-G) Score of 0 or 1 and at Least a 2-grade Improvement From Baseline to Week 16 | Baseline and Week 16
  Percentage of participants achieving a sPGA-G Score of 0 or 1 and at least a 2-grade improvement from baseline to Week 16 will be reported. The sPGA-G is a 6-point scale to assess the severity of genital psoriasis at a given time point. The sPGA-G evaluates erythema, plaque elevation, and scale of genital psoriatic lesions. The severity of genital psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), and very severe (5).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving a Physician's Global Assessment of Hands and Feet (hf-PGA) Score of 0 or 1 and at Least a 2-grade Improvement From Baseline to Week 16 | Baseline and Week 16
  Percentage of participants achieving a hf-PGA score of 0 or 1 and at least a 2-grade improvement from baseline to Week 16 will be reported. The hf-PGA assesses the severity of hand and foot psoriasis using a 5-point scale to score the plaques on the hands and feet as: clear (0), almost clear (1), mild (2), moderate (3), and severe (4).
JNJ-77242113 and Placebo Group: Percent Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) Score at Week 16 | Baseline and Week 16
  Percent change from baseline in mNAPSI score at Week 16 will be reported. The mNAPSI is an index used for assessing and grading the severity of nail psoriasis. Each of the participant's 10 fingernails are evaluated for 7 features. The first 3 features are each scored from 0 to 3 in severity and are (1) onycholysis and oil-drop dyschromia, (2) pitting, and (3) nail plate crumbling. The next 4 features are scored 0 - absent or 1 - present and are (1) leukonychia, (2) splinter hemorrhages, (3) nail bed hyperkeratosis, and (4) red spots in the lunula. The score ranges from 0 to 13 per nail and 0 to 130 for all fingernails.
JNJ-77242113 and Placebo Group: Percent of Participants Achieving Fingernail Physician's Global Assessment (f-PGA) Score of 0 or 1 at Week 16 | Week 16
  Percent of participants achieving f-PGA score of 0 or 1 at Week 16 will be reported. The f-PGA is used to evaluate the current status of a participant's fingernail psoriasis on a scale of 0 to 4 (clear [0], minimal [1], mild [2], moderate [3], or severe [4]).
JNJ-77242113 and Placebo Group: Change From Baseline in PSSD Symptom Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSD symptom score at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Change From Baseline in PSSD Sign Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSD sign score at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants With PSSD Sign Score of 0 at Week 16 | Week 16
  Percentage of participants with PSSD sign score of 0 at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Genital Psoriasis Sexual Frequency Questionnaire (GenPs-SFQ) Item 2 Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving GenPs-SFQ Item 2 score of 0 or 1 at Week 16 will be reported. The GenPs-SFQ is a 2-item participant-reported instrument used to assess the impact of genital psoriasis on the frequency of sexual activity in the last 7 days. Item 1 assesses overall frequency of sexual activity in the last 7 days (none/zero, once, or 2 or more times), and item 2 assesses how frequently genital psoriasis symptoms have limited the frequency of sexual activity in the last 7 days (never [0], rarely [1], sometimes [2], often [3], or always [4]).
JNJ-77242113 and Placebo Group: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving DLQI score of 0 or 1 at Week 16 will be reported. The DLQI is a dermatology specific health-related quality of life (HRQoL) instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Placebo Group: Change From Baseline in Total DLQI Score at Week 16 | Baseline and Week 16
  Change from baseline in total DLQI score at Week 16 will be reported. The DLQI is a dermatology specific HRQoL instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Placebo Group: Change from Baseline in Domain Scores of the Patient-reported Outcomes Measurement Information System-29 (PROMIS-29) Score at Week 16 | Baseline and Week 16
  Change from baseline in domain scores of the PROMIS-29 score at Week 16 will be reported. The PROMIS-29 is a 29-item generic HRQoL survey, assessing each of the 7 PROMIS domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities) with 4 questions for each domain. The questions are ranked on a 5-point Likert scale. There is also a numerical rating scale that ranges from 0 (No pain) to 10 (Worst pain imaginable) for pain intensity. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores on anxiety, depression, fatigue, sleep disturbance, and pain interference indicate more severe symptoms. Higher scores on physical function and social participation indicate better health outcomes.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving DLQI Score of 0 or 1 at Weeks 16 and 24 | Weeks 16 and 24
  Percentage of participants achieving DLQI score of 0 or 1 at Weeks 16 and 24 will be reported. The DLQI is a dermatology specific HRQoL instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
JNJ-77242113 and Deucravacitinib Group: Percentage of Participants Achieving PSSD Symptom Score of 0 at Weeks 16 and 24 | Weeks 16 and 24
  Percentage of participants achieving PSSD symptom score of 0 at Weeks 16 and 24 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Who Achieve PASI 75 Response After Week 24 Among PASI 75 Non-responders to Deucravacitinib at Week 24 | Baseline and from Week 24 through Week 156
  Percentage of participants who achieve PASI 75 response (>=75% improvement in PASI) after Week 24 among PASI 75 Non-responders to deucravacitinib at Week 24 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Who Achieve PASI 90 Response After Week 24 Among PASI 90 Non-responders to Deucravacitinib at Week 24 | Baseline and from Week 24 through Week 156
  Percentage of participants who achieve PASI 90 response (>=90% improvement in PASI) after Week 24 among PASI 90 non-responders to deucravacitinib at Week 24 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving IGA Score of 0 or 1 after Week 24, Among Participants with IGA score >=2 at Week 24 in the Deucravacitinib Group | From Week 24 through Week 156
  Percentage of participants achieving IGA score of 0 or 1 after Week 24, among participants with IGA score >=2 at Week 24 in the deucravacitinib group will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinicaltrial, Study Director — Janssen Research & Development, LLC
Locations (164):
- United States (50):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Integrative Skin Science and Research, Sacramento, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research LLC, Coral Gables, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Hamilton Research LLC, Alpharetta, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - DeNova Research, Chicago, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Northshore Medical Group, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - David Fivenson MD, Dermatology, Ann Arbor, Michigan
  - Michigan Center of Medical Research, Clarkston, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Specialists, Omaha, Nebraska
  - Fife Dermatology, Las Vegas, Nevada
  - StracSkin, Portsmouth, New Hampshire
  - Schweiger Dermatology Group, East Windsor, New Jersey
  - Schweiger Dermatology Group, Hackensack, New Jersey
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Oakview Dermatology, Athens, Ohio
  - Optima Research, Boardman, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Health Concepts, Rapid City, South Dakota
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - National Clinical Research, Richmond, Virginia
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
  - Premier Clinical Research, Spokane, Washington
- Argentina (8):
  - Instituto Medico De Alta Complejidad (IMAC), Buenos Aires
  - ARCIS Salud SRL Aprillus asistencia e investigacion, Buenos Aires
  - Halitus Instituto Medico S.A. - Dermatologia y Estetica, Caba
  - Hospital Italiano de Buenos Aires, Caba
  - Instituto de Neumonologia y Dermatologia, CABA
  - Hospital Italiano de La Plata, La Plata
  - Instituto Caici Srl., Rosario
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Australia (5):
  - North Eastern Health Specialists, Campbelltown
  - Paratus Clinical Research Woden, Canberra
  - Sinclair Dermatology, East Melbourne
  - Skin Health Institute Inc., Melbourne
  - Veracity Clinical Research, Woolloongabba
- Fundacao do ABC Centro Universitario FMABC, Santo André, Brazil
- Canada (8):
  - Enverus Medical, Surrey, British Columbia
  - Karma Clinical Trials Inc., St. John's, Newfoundland and Labrador
  - CCA Medical Research Corporation, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
- Germany (15):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Hautarztpraxis, Bramsche
  - Klinische Forschung Dresden GmbH, Dresden
  - Praxis für Dermatologie und Venerologie, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - MensingDerma research GmbH, Hamburg
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Studienzentrum Dr Schwarz Germany, Langenau
  - Universitatsklinikum Leipzig AOR, Leipzig
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Universitaetsklinikum Mannheim, Mannheim
  - Klinik und Poliklinik fur Dermatologie und Allergologie am Biederstein, München
  - Hautarztpraxis, Potsdam
  - Universitaetsmedizin Rostock, Rostock
- Hungary (8):
  - Pecsi Tudomanyegyetem, Borgyogyaszati Klinika
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Derma-B Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - SZTE AOK Szent-Gyorgyi Albert Klinikai Kozpont, Borgyogyaszati és Allergologiai Klinika, Szeged
  - Allergo-Derm Bakos Kft., Szolnok
  - Medmare Egeszsegugyi Es Szolgaltato Bt., Veszprém
- Japan (23):
  - Fukuoka University Hospital, Fukuoka
  - Hino Dermatology Clinic, Fukutsu
  - Gifu University Hospital, Gifu
  - University of the Ryukyus Hospital, Ginowan
  - Gunma University Hospital, Gunma
  - JR Sapporo Hospital, Hokkaido
  - Asahikawa Medical University Hospital, Hokkaido
  - Tokai University Hospital, Isehara
  - Teikyo University Hospital, Itabashi Ku
  - St Marianna University Hospital, Kawasaki
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu-shi
  - Nagoya City University Hospital, Nagoya
  - Kume Clinic, Nishiku
  - Takagi Dermatological Clinic, Obihiro Shi
  - Public Interest Incorporated Foundation Nipoon Life Saiseikai Nippon Life Hospital, Osaka
  - Kindai University Hospital, Sakai
  - Sapporo Skin Clinic, Sapporo
  - Tohoku University Hospital, Sendai
  - The University of Osaka Hospital, Suita
  - Jitaikai Tachikawa dermatology clinic, Tachikawa
  - Shirasaki Dermatology Clinic, Takaoka Shi
  - Tokyo Medical University Hospital, Tokyo
  - Mie University Hospital, Tsu
- Poland (16):
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - Specderm Poznanska sp j, Bialystok
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Medyczne dr Rajzer Sp z o o, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Medyczne Promed, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski S C, Osielsko
  - SOLUMED Centrum Medyczne, Poznan
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - Dorota Bystrzanowska High-Med. Przychodnia Specjalistyczna, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - DERMMEDICA Sp.z o.o., Wroclaw
  - Wro Medica, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
- Spain (12):
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Grupo Dermatologico Y Estetico Pedro Jaen, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia
- Taiwan (7):
  - Chang Kung Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (4):
  - Guys and St Thomas NHS Foundation Trust, London
  - Royal Berkshire Hospital, Reading
  - Salford Royal Hospital, Salford
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gold LS, Armstrong AW, Bissonnette R, Magnolo N, Vender RB, Sebastian M, Galimberti ML, Tsianakas A, Arnone M, Wallace P, Simon M, Riera-Monroig J, Gerdes S, Waibel J, Gonzalez-Cantero A, Schwarz B, Tada Y, Cecchini M, Ehst B, Kircik L, Kephart L, Reyes-Servin O, Edem BE, Campbell JH, Shen YK, Cresswell K, Li S, DeKlotz CMC, Nunes F, Papp KA. Once-daily oral icotrokinra versus placebo and once-daily oral deucravacitinib in participants with moderate-to-severe plaque psoriasis (ICONIC-ADVANCE 1 & 2): two phase 3, randomised, placebo-controlled and active-comparator-controlled trials. Lancet. 2025 Sep 27;406(10510):1363-1374. doi: 10.1016/S0140-6736(25)01576-4. Epub 2025 Sep 18. PMID 40976249